CLINICAL TRIAL: NCT02939469
Title: STTR Phase II : Skin Sympathetic Nerve Activity and Cardiac Arrhythmias
Brief Title: Skin Sympathetic Nerve Activity and Cardiac Arrhythmias
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The PI passed away.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Florian Rader, Co-Director, Clinic for Hypertrophic Cardiomyopathy and Aortopathies, Smidt Heart Institute, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro 42959
Record Dates: First submitted 2016-10-11; First posted 2016-10-20 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Sympathetic Nerve Activity
Keywords: Sympathetic Nerve Activity; Skin Sympathetic Nerve Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: Sympathetic nerve activity (Experimental): Healthy volunteers will undergo microneurography, and non invasive sympathetic nerve activity by EKG analysis at baseline and in response to stress.
  Interventions: Other: Physiologic maneuvers

INTERVENTIONS:
Other: Physiologic maneuvers — Subjects will perform
  Valsalva maneuver Hand Grip Post exercise cuff occlusion Loud Noise and Skin pinch

SUMMARY:
Since the invention of electrocardiogram (ECG), ECG has been an important part of clinical practice. A primary reason for the popularity of the ECG is that it is non-invasive and can be performed in any patient by placing electrodes on the skin. The present methods of ECG recording focus on detecting electrical signals from the heart. the investigators propose that with high frequency sampling and high pass filtering, the investigators can also record SNA from the skin. The somata of the subcutaneous sympathetic nerves on the skin are located at the ipsilateral cervical and stellate ganglia. Because the left stellate ganglion nerve activity (SGNA) is known to trigger cardiac arrhythmias, including AF, VF and VF, It is possible that skin SNA can also be used for arrhythmia prediction. the investigators tested that hypothesis in our preclinical studies (supported by R01 HL71140) using canine models. The results showed that subcutaneous nerve activity (SCNA) recorded with implanted electrodes can be used to estimate stellate ganglion nerve activity(SGNA) in normal dogs and in a canine model of ventricular arrhythmia and sudden death. the investigators also showed that SCNA is more accurate than heart rate variability in estimating cardiac sympathetic tone in ambulatory dogs with myocardial infarction.Therefore, SKNA and SCNA may be useful in estimating cardiac sympathetic tone. In addition to studying the autonomic mechanisms of cardiac arrhythmia, these new methods may have broad application in studying both cardiac and non-cardiac diseases. For example, sympathetic tone is important in the pathogenesis of heart failure, atherosclerosis, peripheral neuropathies, epilepsy, vasovagal syncope, renal failure, hypertension and many others diseases. Direct SKNA and SCNA recording may provide new approaches to study the mechanisms of these common diseases. SKNA recording may also have immediate clinical applications by assisting in the diagnosis and treatment of hyperhidrosis (sweaty palms), paralysis, stroke, diabetes, and neuromuscular diseases. It may be used to assist biofeedback monitoring performed by neurologists to control neuropsychiatric disorders. Because of these potential clinical and commercial applications, the investigators propose that this research project is significant.

b. Innovation

* Using conventional electrodes on the skin to record SNA. The neuECG utilizes the conventional skin electrodes that are widely used in health care facilities. Skin SNA had been recorded using microneurography techniques, and had been estimated using cutaneous blood flow (vasodilator responses) skin temperature, skin conductance and sweat release. However, microneurography cannot be used in ambulatory patients. The other methods are not direct measurements of SNA. neuECG is the first method that can directly and non-invasively measure the SNA from the skin.
* Automated real-time signal processing. the investigators will develop signal processing software to automatically eliminate noise, such as that generated by muscle contraction, electrical appliances, body motion, respiration, and radiofrequency signals. The remaining signals are then processed to separately display in real time to provide health care providers a new method to instantly estimate sympathetic tone. The ECG signals are used for automated arrhythmia detection while the SNA signals are available for risk stratification. This approach allows us to improve and broaden the clinical application of Einthoven's original invention by simultaneous detecting ECG and SNA from the skin.
* SKNA patterns as new biomarkers. the investigators have identified unique SKNA patterns that precede the onset of human AF. If proven correct by Specific Aim 3, this new biomarker can help physicians to estimate the arrhythmia risk and to predict the efficacy of catheter ablation for AF.

DETAILED DESCRIPTION:
Background Cardiac sympathetic innervation comes from the paravertebral cervical and thoracic ganglia. Among them, the stellate (cervicothoracic) ganglion is a major source of sympathetic innervation. It constantly connects with phrenic nerves and almost as often to the vagal nerves.37 The paravertebral ganglia also directly connect with spinal nerves, which connect with the intercostal nerves. These intercostal nerves split into ramus cutaneous lateralis and a deep branch to the musculus rectus abdominis. Histological studies of human skin biopsy confirmed the presence of abundant sympathetic nerves in arteriovenous anastomoses arrector pilorum muscles, and arterioles. Using horseradish peroxidase as tracer, Baron et al and Taniguchi et al found that all skin sensory and sympathetic neurons are located ipsilaterally. The sympathetic somata are located in the middle cervical and stellate ganglia as well as the thoracic ganglia. Because of the direct and extensive connections among various nerve structures, it is possible for the sympathetic nerves in the various structures to activate simultaneously. Therefore, the investigators hypothesized that SKNA recorded from the upper thorax can be used to estimate the cardiac sympathetic tone.

Utilize the differential frequency contents of ECG and SNA to record neuECG To preserve the signal and eliminate noise, the American Heart Association (AHA) standard recommendation for low pass filtering of the ECG is 150 Hz for adolescents and adults, and 250 Hz for children. Higher frequency signals, although known to be clinically important, are routinely eliminated by this low pass filtering. Because there is no need to record high frequency signals, the conventional ECG and Holter monitoring devices do not have a wide bandwidth and high sampling rate. neuECG recording takes a different approach. the investigators use equipment with wide bandwidth (2K Hz) and high sampling rate (4K/s-10K/s) to record the signals from the skin. The signal is then band passed between 0.5 Hz and 150 Hz to display ECG signal. The same signals are then high passed at > 150 Hz to reveal nerve activities. Figure 1 illustrates the above concept. It shows Fast Fourier Transform (FFT) analyses of the signals recorded from the skin. High pass filtering at 150 Hz eliminated the ECG signals. The remaining high frequency signals may contain both muscle and nerve activities. McAuley et al reported that the electromyography (EMG) usually has a frequency of <100 Hz. At most, small amounts of muscle activities could reach 400 Hz. By high pass filtering at 500 Hz, the EMG is eliminated but so are other signals with frequencies < 500 Hz. The standard high pass setting for microneurography study is 700 Hz. High pass filtering at 500 or 700 Hz increased the specificity but reduced the sensitivity of SKNA recording. The signal to noise ratio is reduced. However, the basic patterns of nerve discharges remain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years of age
* BMI < 35 kg/m2

Exclusion Criteria:

* History of hypertension, diabetes, pulmonary disease, metabolic disease or heart failure
* Cardiac rhythm disorder, specifically: rhythm other than sinus
* Use of any medications other than common supplements
* Unable to perform handgrip exercise
* Pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Chane in Sympathetic nerve activity | Change from baseline in sympathetic nerve activity at 2 hours
  Multi-unit recordings of sympathetic nerve activity will be obtained with single-use sterile

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States